CLINICAL TRIAL: NCT02541500
Title: An Open-label Study of Oral Minocycline for the Treatment of Patients With Co-occurring Opioid and Amphetamine-type Stimulant Dependence (COATS)
Brief Title: An Open Label Study of Oral Minocycline for the Treatment of Patients With Co-occurring Opioid and ATS Dependence
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiti Sains Malaysia (Other)
Collaborators: Yale University (Other)
Responsible Party: Principal Investigator, Vicknasingam B Kasinather, Dr, Universiti Sains Malaysia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00004494
Record Dates: First submitted 2015-06-29; First posted 2015-09-04 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-09

CONDITIONS: Heroin Dependence; Amphetamine Dependence
Keywords: minocycline; amphetamine type stimulant dependence
MeSH Terms: conditions — Heroin Dependence; Amphetamine-Related Disorders; cyclopia sequence | interventions — Minocycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Minocycline (Experimental): Patients in this arm will receive oral minocycline
  Interventions: Drug: Minocycline

INTERVENTIONS:
Drug: Minocycline — Oral minocycline 200 mg daily will be started on day six of treatment for a period of four months
  Other Names: Borymycin

SUMMARY:
The proposed study will evaluate the tolerability, acceptability and potential efficacy of minocycline for the treatment of co-occurring opioid and amphetamine-type stimulant (ATS) dependence. In the proposed clinical trial, all patients will first discontinue illicit opioid and ATS and be inducted onto buprenorphine maintenance treatment (BMT) in the inpatient ward at the department of psychiatry before beginning to receive minocycline. Tolerability and acceptability will be evaluated by assessing the rates of patient retention during treatment, patient satisfaction with treatment and adverse effects during treatment. The potential efficacy of minocycline will be evaluated with regard to the primary outcome measure: reductions in ATS use , based on urine toxicology testing and self-report. Secondary outcome measures include retention, reduction in HIV risk behaviors and improvements in functional status.

DETAILED DESCRIPTION:
Additional data available to this project will come from contemporaneous and historical drug treatment clinical trials and treatment programs conducted at HUSM with similar populations of patients and proposed/described as other components of the cluster of research projects described in the overall Research University Team Grant proposal. Comparisons of treatment process and outcome measures collected in this proposed clinical trial with data collected in contemporaneous and historical controls will enhance our ability to evaluate the potential efficacy of minocycline as treatment agent for co-occurring opioid and amphetamine-type stimulant (ATS) dependence. Data from patients receiving other drug treatments at HUSM will be used as reference points to evaluate potential effect sizes of treatment effects associated with minocycline treatment. The preliminary data on treatment retention data, patient satisfaction, potential adverse effects, and efficacy will be used as preliminary/pilot research when designing and applying for funding support for future large scale randomized clinical trials aimed at the development of effective medically based treatments of opiate and ATS abuse or dependence.

Over the past decade, amphetamine-type stimulant (ATS) has also emerged as a major drug problem. Globally, ATS is now the second most commonly used illicit drug type and is more widely used than heroin. ATS abuse is especially prevalent and problematic in the Asian region, where ATS production, use, drug seizures, and demand for treatment have continued to increase. Injection of methamphetamine has been reported in Malaysia (Chawarski et al, 2006) and other south-east Asian countries (McKetin, 2008). In the most recent survey of out-of-treatment heroin IVDU in cities across Malaysia, more than 60% report current ATS use, and 29% inject ATS (Chawarski et al, 2012).

ATS use is associated with increased HIV transmission behavioral risks. The connection of heroin, methamphetamine and HIV in Malaysia is well documented (Chawarski et al, 2006). Increased needle sharing and risky sexual behaviors lead to increased prevalence of HIV infection. ATS use exacerbates HIV transmission risk through a number of mechanisms: ATS users report engaging in more frequent and more risky sexual behaviors while using ATS and in more frequent needle sharing. ATS is also associated with impairments of mood and executive functioning that may persist for prolonged periods and may contribute to relapse to drug use, thus all other problems.

Drug abuse has been a major problem in Kelantan for the past several decades (Suarn & NorAdam,1993) and ATS has been gaining momentum over the past decade. The number of individuals arrested annually for ATS in Kelantan increased over the past 5 years from 2900 in 2007 to 5300 in 2010. For the past 5 years, Kelantan has also led Malaysia in having the highest population prevalence of HIV infection, at 47 per 100,000 in 2008, nearly 4 times the prevalence reported for the rest of Malaysia. Kelantan also has the highest number of women with HIV in Malaysia with more than 1200 reported in 2008, suggesting that HIV is making the transition to the general population. A large proportion of treatment seeking drug users in Kelantan are HIV positives and are susceptible to high mortality (JKNK, 2012).

Minocycline is a broad-spectrum antibiotic derived from tetracycline. Minocycline is substantially more lipid-soluble than other tetracyclines, thus minocycline readily crosses the blood-brain barrier, and its potential efficacy for treating ATS dependence derives from its effects on dopamine on glutamate neurotransmission in the brain and its anti-inflammatory, neuro-protective and cognitive-enhancing effects in the brain (Dean et al, 2012). Glutamate along with dopamine plays a key role in the rewarding and addictive effects of amphetamine, methamphetamine, and other stimulants. Input from glutamatergic pathways in brain reward centers enhances dopaminergic transmission in these pathways and reward. Blockade of glutamate receptors in these regions prevents many of the behavioral effects of ATS or other stimulants and prevents reinstatement of stimulant use in animal studies. Glutamate plays a key role in learning and memory, and blockade of glutamate interferes with consolidation of memory for the rewarding effects of stimulants.

Minocycline, one of the very few medications affecting glutamate transmission, attenuates many of the behavioral effects of stimulants in animal models, attenuates release of dopamine in brain reward pathways in response to stimulants. It has cognitive-enhancing effects in humans, and improves stimulant-induced and phencyclidine-induced cognitive impairments. In animal models, minocycline improved stimulant-induced or phencyclidine-induced impairments of object recognition, sensorimotor gating, and visuospatial memory. A study of nicotine addiction showed greater reduction in craving for cigarettes while on minocycline as compared to placebo (Sofuoglu et al, 2009).

In another study (Sofuoglu et al, 2011), minocycline attenuated the subjective, rewarding effects of amphetamine administration in healthy human volunteers, reduced plasma cortisol levels following amphetamine administration, and improved reaction times on a cognitive performance task testing attention. The cognitive-enhancing effects of minocycline have been found in individuals with schizophrenia, who showed improved working memory, cognitive flexibility and cognitive planning in response to minocycline. Addition of minocycline early in the treatment improves negative symptoms in patient with schizophrenia (Chaudry et al, 2012).Minocycline exerts neuroprotective effects but under certain circumstances, also have neurotoxic consequences (Plane et al, 2010). Reserchers in Japan reported a case of a female patient whose psychotic symptoms in methamphetamine use disorder were successfully improved by minocycline, even though the precise mechanisms were not understood then (Tanibuchi et al, 2010).

Very rarely, minocycline is associated with some severe problems, including colitis, infection with non-susceptible organisms, liver damage, (MacNeil et al,1997), benign intracranial hypertension, skin rashes, autoimmune disorders or allergic reactions. Although these problems occur very rarely, we plan to monitor patients for adverse effects closely throughout the study to ensure early detection and prompt treatment of any serious advere effect, if one should occur. Additionally, patients treated for acne with minocycline may be treated with minocycline for many years, while in the proposed study we are planning to treat patients with minocycline for a very limited period, 4 months. We anticipate that, if it is found to be efficacious for treating ATS abuse or dependence, minocycline would be used in the initial phase of treatment to help patients consolidate a period of abstinence from ATS and develop healthy, drug-free life styles; we do not anticipate that minocycline would be used for the long-term maintenance treatment of ATS abuse or dependence.

In addition to detoxification and treatment medications, a manual-guided educational drug and HIV risk reduction counseling (EDRC) will be provided to all participants. EDRC provides education about medical understanding of opioid and ATS addiction, highly effective strategies used in successful drug recovery efforts, medical and other harmful consequences of drug use includingHIV and other infectious disease transmission, as well as about effective prevention of all negative consequences of illicit drug use (Chawarski et al, 2008). It helps patient to remain in treatment, adhere to prescribed medications, abstain from or reduce illicit opioid and ATS use and HIV risk behaviors, and make life-style changes fostering sustained recovery. It also teaches basic cognitive and behavioral coping skills that increase the patients' chances to reach sustained and prolonged recovery from drugs. For HIV positive patients, EDRC encourages patients to attend the HIV clinic and adhere to monitoring, medication, and other treatment recommendations. EDRC will be provided by trained and supervised nursing personnel, drug counselors, or therapists. It will be offered in individual format with the frequency ranging from 3 times per week during detoxification to once per week during the outpatient phase of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Meet DSM-IV criteria for both opioid and ATS dependence, as assessed by the Structured Clinical Interview for DSM (SCID)
2. ActiveCOATS dependence as documented by ATS and opioid-positive urine tests and a report of at least 2 or more days per week of ATS use over the past month.
3. Age 18 - 65 years old

Exclusion Criteria:

1. Liver enzymes greater than 3 times the upper limit of normal or evidence of liver failure or acute hepatitis.
2. Having serious medical or psychiatric illnesses: (including current psychotic disorder, major depression, suicidal or homicidal ideations) or taking medications to treat depression or psychosis.
3. Refused informed consent or inability to understand the protocol or assessment questions.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-04; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in illicit ATS use, | 18 weeks
  This will be measured from baseline over time during treatment based on urine toxicology testing and self-report

SECONDARY OUTCOMES:
Reductions in sexual and drug-related HIV risk behaviors | 18 weeks
  Measured by repeated assessments of sexual and HIV risk behaviors during treatment
Measure improvements in neuropsychological functioning | 18 weeks
  Measured by repeated assessments of neuropsychological functioning

CONTACTS AND LOCATIONS:
Overall Officials: Imran Ahmad, MBBS, Principal Investigator — University Science Malaysia
Locations (1):
- University Science Malaysia, Kota Bharu, Kelantan, Malaysia